CLINICAL TRIAL: NCT01232504
Title: Effect of Granulocyte-macrophage Stimulating Factor on Prevention and Treatment of Invasive Fungal Diseases in the Recipients of Allogeneic Stem Cell Transplantation: A Prospective Multicenter Randomized Phase 4 Trial
Brief Title: Antifugal Effect of Recombinant Human Granulocyte-macrophage Stimulating Factor (rhGM-CSF) in Patients Post Allo-HSCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Shanghai Jiao Tong University Affiliated First People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: L-09-01
Record Dates: First submitted 2010-10-25; First posted 2010-11-02 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Mycoses
Keywords: Allo-HSCT; rhGM-CSF; Systemic fungal infection (SFI)
MeSH Terms: conditions — Mycoses | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rhGM-CSF group (Experimental): subcutaneous 5-7μg/kg/d Recombinant Human Granulocyte-macrophage Stimulating Factor (rhGM-CSF) once daily
  Interventions: Drug: rhGM-CSF group
- rhG-CSF+rhGM-CSF group (Active Comparator): a combination of 2-3μg/kg/d Recombinant Human Granulocyte-macrophage Stimulating Factor (rhGM-CSF) and 2-3μg/kg/d Recombinant Human Granulocyte Stimulating Factor (rhG-CSF) each
  Interventions: Drug: rhG-CSF+rhGM-CSF group
- rhG-CSF group (Active Comparator): subcutaneous 5-7μg/kg/d Recombinant Human Granulocyte Stimulating Factor (rhG-CSF) once daily
  Interventions: Drug: rhG-CSF group

INTERVENTIONS:
Drug: rhGM-CSF group — subcutaneous rhGM-CSF 5-7μg/kg/d , started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
  Other Names: Topleucon®; Granulocyte Macrophage Colony Stimulating Factor
  Arms: rhGM-CSF group
Drug: rhG-CSF+rhGM-CSF group — a combination of 2-3μg/kg/d rhGM-CSF and 2-3μg/kg/d rhG-CSF each after transplantation, started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
  Other Names: Topleucon®; Granulocyte Macrophage Colony Stimulating Factor; Granulocyte Colony Stimulating Factor
  Arms: rhG-CSF+rhGM-CSF group
Drug: rhG-CSF group — subcutaneous rhGM-CSF 5-7μg/kg/d , started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
  Other Names: Granulocyte Colony Stimulating Factor; Topleucon®
  Arms: rhG-CSF group

SUMMARY:
We conducted a prospective, multicenter, open-label randomized trial to compare the antifungal effect of Recombinant Human Granulocyte-macrophage Stimulating Factor (rhGM-CSF), Recombinant Human Granulocyte Stimulating Factor (rhG-CSF) or a combination of rhGM-CSF and rhG-CSF for neutropenic patients undergoing allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
From Sept 2009 to Dec 2012, we recruited consecutive patients with hematological diseases undergoing allogeneic stem cell transplantation at 5 institutions in China. Recipients between ages of 14 to 60 years old were eligible. Eligible patients were randomized to receive once daily subcutaneous 5-7μg/kg/d GM-CSF (Molgramostim, TOPLEUCON®; Xiamen Amoytop Biotech Co., Ltd., China) (GM-CSF group), 5-7μg/kg/d G-CSF (G-CSF group), or a combination of 2-3μg/kg/d GM-CSF and 2-3μg/kg/d G-CSF each (G-CSF+GM-CSF group). Administration of CSFs was started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days). If absolute neutrophil count (ANC) decreased to < 1.5×10(9)/L within 5 days after withdrawal of CSFs, the same CSF would be resumed until the absolute neutrophil count (ANC) reached 1.5×10(9)/L again. All patients received antimicrobial prophylaxis with oral levofloxacin 500 mg daily and antifungal prophylaxis with oral fluconazole 200 mg daily.

ELIGIBILITY:
Inclusion Criteria:

* Age 14~60 years old
* Allogenic hematological stem cell transplantation(HSCT) patients.
* Cardiac ejection factor ≥ normal upper limit, Aspartate aminotransferase and/or Alanine aminotransferase < 2 upper limit of normal, and/or total bilirubin < 2.5 upper limit of normal, creatinine < upper limit of normal.
* Informed consent.

Exclusion Criteria:

* Evidence of proven, probable or possible fungal infection at the time of enrollment.
* Patients were receiving anti-fungal treatment with proven SFI before transplantation.
* A history of hypersensitivity to G-CSF or GM-CSF.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2009-09; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wang, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (5):
- China (5):
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Tongji Hospital, Wuhan, Hubei
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

REFERENCES:
- [Derived] Wan L, Zhang Y, Lai Y, Jiang M, Song Y, Zhou J, Zhang Z, Duan X, Fu Y, Liao L, Wang C. Effect of Granulocyte-Macrophage Colony-Stimulating Factor on Prevention and Treatment of Invasive Fungal Disease in Recipients of Allogeneic Stem-Cell Transplantation: A Prospective Multicenter Randomized Phase IV Trial. J Clin Oncol. 2015 Dec 1;33(34):3999-4006. doi: 10.1200/JCO.2014.60.5121. Epub 2015 Sep 21. PMID 26392095

RESULTS

PARTICIPANT FLOW:
Groups:
- rhGM-CSF Group: subcutaneous recombinant human granulocyte-macrophage stimulating factor (rhGM-CSF) 5-7μg/kg/d , started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
- rhG-CSF+ rhGM-CSF Group: a combination of 2-3μg/kg/d recombinant human granulocyte-macrophage stimulating factor (rhGM-CSF) and 2-3μg/kg/d recombinant human granulocyte stimulating factor (rhG-CSF) each after transplantation, started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
- rhG-CSF Group: subcutaneous recombinant human granulocyte stimulating factor (rhGM-CSF) 5-7μg/kg/d , started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
Period: Overall Study
Arm/Group | rhGM-CSF Group | rhG-CSF+ rhGM-CSF Group | rhG-CSF Group
Started | 68 | 69 | 69
Completed | 59 | 67 | 61
Not Completed | 9 | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- rhG-CSF+ rhGM-CSF Group: a combination of 2-3μg/kg/d rhGM-CSF and 2-3μg/kg/d rhG-CSF each after transplantation, started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
- rhG-CSF Group: subcutaneous rhG-CSF 5-7μg/kg/d , started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
- Total: Total of all reporting groups
Arm/Group | rhGM-CSF Group | rhG-CSF+ rhGM-CSF Group | rhG-CSF Group | Total
Number analyzed (Participants) | 68 | 69 | 69 | 206
Age, Continuous [Median (Full Range); unit: years] | 30.68 [14 to 60] | 32.55 [14 to 56] | 32.04 [15 to 53] | 31.75 [14 to 60]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 5 | 9 | 22
  Between 18 and 65 years | 60 | 64 | 60 | 184
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 32 | 25 | 74
  Male | 51 | 37 | 44 | 132
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 68 | 69 | 69 | 206
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 68 | 69 | 69 | 206

OUTCOME MEASURES:

1. Secondary Outcome: Hematological Engraftment
Description: The median time of neutrophil and platelet recovery .
Time Frame: 100 days post transplant
Population: The number of intention-to-treat patients is 206. The hematological engraftment analysis within 100 day is based on intention-to-treat (ITT)patients .
Measure: Median (Full Range); unit: days
Groups:
- rhG-CSF + rhGM-CSF Group: a combination of 2-3μg/kg/d rhGM-CSF and 2-3μg/kg/d rhG-CSF each after transplantation, started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
Arm/Group | rhGM-CSF Group | rhG-CSF + rhGM-CSF Group | rhG-CSF Group
Number analyzed (Participants) | 68 | 69 | 69
days
  Median time for neutrophil recovery to 0.5×10(9)/L | 13 [9 to 25] | 11 [5 to 28] | 11 [6 to 28]
  Median time for platelet recovery to 50 × 10(9)/L | 18 [10 to 200] | 19 [10 to 200] | 25 [12 to 200]

2. Secondary Outcome: Transplant Related Mortality
Description: Transplant related mortality within 100 days after Allogeneic Stem Cell Transplantation (Allo-HSCT).
Time Frame: 100 days post transplant
Population: The number of intention-to-treat patients is 206. The transplant related mortality analysis within 100 day is based on intention-to-treat (ITT) patients .
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rhGM-CSF Group | rhG-CSF+ rhGM-CSF Group | rhG-CSF Group
Number analyzed (Participants) | 68 | 69 | 69
percentage of participants | 8.8 [3.3 to 18.2] | 8.7 [3.3 to 17.9] | 21.7 [12.7 to 33.3]

3. Secondary Outcome: Incidence of Ⅱ- Ⅳ Acute Graft Versus Host Disease (aGVHD)
Description: Incidence of Ⅱ- Ⅳacute graft versus host disease (aGVHD) within 100 days after allogeneic stem cell transplantation (Allo-HSCT).The severity of acute GVHD in the three main target organs (skin, liver, gastrointestinal tract) was assigned stage 1 to 4 based on accepted criteria (Consensus Conference on Acute GVHD Grading).
Time Frame: 100 days post transplant
Population: The number of intention-to-treat patients is 206. The incidence of aGVHD analysis is based on intention-to-treat (ITT) patients .
Measure: Number (95% Confidence Interval); unit: percentage of partipants
Groups:
- rhGM-CSF: 5-7μg/kg per day
  rhGM-CSF: 5-7μg/kg daily subcutaneously（sc）without interruption until neutrophils≥1.5×10(9)/L for two continuous days,starting 5 days after transplantation.
- rhGM-CSF Plus rhG-CSF: rhGM-CSF and rhG-CSF both at 2-3μg/kg per day
  rhGM-CSF plus rhG-CSF: rhGM-CSF and rhG-CSF (both at 2-3μg/kg/d) subcutaneously（sc）without interruption until neutrophils≥1.5×10(9)/L for two continuous days,starting 5 days after transplantation.
- rhG-CSF: 5-7μg/kg per day
  rhG-CSF: 5-7μg/kg daily subcutaneously（sc）without interruption until neutrophils≥1.5×10(9)/L for two continuous days,starting 5 days after transplantation.
Arm/Group | rhGM-CSF | rhGM-CSF Plus rhG-CSF | rhG-CSF
Number analyzed (Participants) | 68 | 69 | 69
percentage of partipants | 30.88 [20.2 to 43.3] | 24.64 [15.1 to 36.5] | 21.74 [12.7 to 33.3]

4. Primary Outcome: Incidences of Invasive Fungal Diseases (IFD)
Description: The incidence of proven and probable Invasive fungal diseases (IFD) within 100 days post transplantation
Time Frame: 100 day post transplant
Population: The number of intention-to-treat patients is 206. The incidence of invasive fungal infection analysis within 100 day is based on intention-to-treat (ITT)patients .
Measure: Number; unit: percentage of partipants
Groups:
- rhG-CSF+ rhGM-CSF: a combination of 2-3μg/kg/d rhGM-CSF and 2-3μg/kg/d rhG-CSF each after transplantation, started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
Arm/Group | rhGM-CSF Group | rhG-CSF+ rhGM-CSF | rhG-CSF Group
Number analyzed (Participants) | 68 | 69 | 69
percentage of partipants | 11.76 | 10.14 | 23.19

5. Secondary Outcome: IFD Related Mortality
Description: IFD-related mortalities after a median follow-up of 600 days.
Time Frame: 3-1099 days
Population: The number of intention-to-treat patients is 206. The IFD related mortality analysis is based on intention-to-treat (ITT) patients .
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- rhGM-CSF+ rhG-CSF Group: a combination of 2-3μg/kg/d rhGM-CSF and 2-3μg/kg/d rhG-CSF each after transplantation, started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
- rhG-CSFgroup: subcutaneous rhG-CSF 5-7μg/kg/d , started on day 5 post-transplant and continued until recovery from neutropenia (absolute neutrophil count [ANC] > 1.5×10(9)/L for 2 consecutive days).
Arm/Group | rhGM-CSF Group | rhGM-CSF+ rhG-CSF Group | rhG-CSFgroup
Number analyzed (Participants) | 68 | 69 | 69
percentage of participants | 1.47 [0.04 to 7.92] | 1.45 [0.04 to 7.81] | 11.59 [5.14 to 21.57]

6. Secondary Outcome: Relapse Related Mortality
Description: Relapse related mortality after a median follow-up of 600 days.
Time Frame: 3～1099 days
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | rhGM-CSF Group | rhGM-CSF+ rhG-CSF Group | rhG-CSFgroup
Number analyzed (Participants) | 68 | 69 | 69
percentage of participants | 5.8 | 8.7 | 4.35

7. Secondary Outcome: Graft Versus Host Disease (aGVHD) Related Mortality
Description: Graft versus host disease (aGVHD) related mortality after a median follow-up of 600 days .
Time Frame: 3-1099 days
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | rhGM-CSF Group | rhGM-CSF+ rhG-CSF Group | rhG-CSFgroup
Number analyzed (Participants) | 68 | 69 | 69
percentage of participants | 8.82 | 4.35 | 7.25

8. Secondary Outcome: Hemorrhage Related Mortality
Description: Hemorrhage related mortality after a median follow-up of 600 days
Time Frame: 3-1099 days
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | rhGM-CSF Group | rhGM-CSF+ rhG-CSF Group | rhG-CSFgroup
Number analyzed (Participants) | 68 | 69 | 69
percentage of participants | 5.88 | 1.45 | 1.45

9. Secondary Outcome: Infection Related Mortality
Description: Infection related mortality after a median follow-up of 600 days.
Time Frame: 3～1099 days)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | rhGM-CSF Group | rhGM-CSF+ rhG-CSF Group | rhG-CSFgroup
Number analyzed (Participants) | 68 | 69 | 69
percentage of participants | 1.47 | 5.8 | 14.50

ADVERSE EVENTS:
Time Frame: 28 days post transplant
Arm/Group | rhGM-CSF Group | rhG-CSF + rhGM-CSF Group | rhG-CSF Group
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/69 | 0/69
Other Adverse Events (participants affected / at risk) | 32/68 | 31/69 | 28/69
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rhGM-CSF Group (N=68) | rhG-CSF + rhGM-CSF Group (N=69) | rhG-CSF Group (N=69)
fever (Infections and infestations) | 32 | 31 | 28

LIMITATIONS AND CAVEATS:
The limitations of the current study included the lack of blinding and placebo group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No